CLINICAL TRIAL: NCT01427894
Title: The Combined Effects of Maternal Singing During Skin to Skin Contact (Kangaroo Care) in Preterm Infants in the Neonatal Intensive Care Unit Environment.
Brief Title: Maternal Singing During Kangaroo Care in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mc(0023)(2011)ctil
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2011-09

CONDITIONS: Prematurity; Maternal Anxiety
Keywords: Prematurity; Music; Kangaroo Care; Bonding Mother infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maternal Singing (Experimental): Maternal singing during Kangaroo Care of stable preterm infants
  Interventions: Other: Maternal singing with Kangaroo Care
- Kangaroo Care (No Intervention): Kangaroo Care without singing

INTERVENTIONS:
Other: Maternal singing with Kangaroo Care — Maternal singing with Kangaroo Care
  Arms: Maternal Singing

SUMMARY:
Study objective is to evaluate the additive effect of maternal singing during skin to skin contact (Kangaroo Care) on anxiety reduction both to infants and their mothers.

DETAILED DESCRIPTION:
Maternal singing to preterm infants during Kangaroo Care intervention, is it beneficial?

Protocol

Maternal voice is a predominant source of multimodal stimulation for the developing fetus that is largely lost for the preterm infant amidst the unfiltered levels of auditory stimuli in the neonatal intensive care unit (NICU). These elevated levels of auditory stimulation in the NICU can interfere with an infant's sleep and have a negative effect on vital signs and oxygen saturation. Common sources of sound for the preterm infant are derived from routine incubator noise, monitoring alarms, and the speech sounds of healthcare team, all of which they would not typically encounter if life in the uterus had continued to term. In the midst of these additional sounds, preterm infants lose significant contact with an auditory stimulus they would typically be exposed to until full-term birth (their mothers' voice).

Skin to skin contact care (Kangaroo care) was found to produce cardiorespiratory stability, decrease apneic and periodic breathing, and improve sleep patterns and weight gain in preterm infants. This technique has also been shown to help mothers of preterm infants to develop and strengthen self-confidence and attachment behaviors, leading to reduced stress response. Live music was shown to have a beneficial effect on psychophysiological responses in both mothers and preterm infants during their stay in the NICU.

Aim: To evaluate the combined influence of live maternal singing during kangaroo care (KC) on maternal anxiety and stable preterm infants' responses.

Participants

Inclusion criteria clinically stable infants

postmenstrual age <37 weeks

normal hearing confirmed by measurement of distortion product otoacoustic emission (DPOAE).

Exclusion criteria

observed hyperresponsiveness to live music

congenital anomaly that mainly affects hearing

medication intake (phenobarbital, furosemide, gentamycin) that might interfere with the reaction to musical stimuli

brain anomalies associated with neurological disorders (grade 3-4 intraventricular hemorrhage, periventricular leukomalacia).

Maternal inclusion criteria

ability to hear

literary ability to read and answer an anxiety questionnaire

Maternal exclusion criteria

signs or medical history of postpartum depression.

Procedure A within-subject, crossover, repeated design will be used with participants acting as their own controls. Before starting the research, mothers will get a professional guidance of singing lullabies to their offspring, by a music therapist (E.G). The mothers will be sitting at the infants' bedside and the child will be placed in the kangaroo position with skin-to-skin contact with the mother. Each therapy session will start 30 minutes after feeding to get a relaxed infant and to test the intervention with no disturbances such as hunger. As recommended the infants will receive either KC alone for 30 minutes or KC combined with maternal singing for 30 minutes. According to the randomization schedule, both therapies will be performed in the afternoon after finishing the medical and nursing rounds, in alternating order 3 to 5 days apart to allow for a washout period, and included the same music. Monitor alarms will be silence and the door closed.

Objective Sound Measurements Music and background sound levels will be checked 10 cm from the infant's ear with a sound analyzer and a decibel scale filter (407790 Octave Band Sound Analyzer, type 2 Integrating Sound Level Meter and Decibel-A Scale Filter, respectively; Extech Instruments, Melrose, MA, USA).

Infant and Maternal Measures For accuracy, neonatal and maternal heart rates, oxygen saturation levels, and respiratory rates will be recorded continuously and documented every 2 minutes during all sessions. A 7-point scale to assess infants' behavioral state (deep sleep, light sleep, drowsy, quiet awake or alert, actively awake and aroused highly aroused, upset, or crying, and prolonged respiratory pause > 8 seconds) and a self-report questionnaire comprising 20 descriptive statements for measuring maternal anxiety symptoms (state-trait anxiety inventory [STAI] scale will be used at the beginning and the end of each intervention. Higher scores indicate greater anxiety, with a possible score of 20 to 80 points. Additional maternal measures will be age, ethnicity (Arab/Jews), education (8 years, elementary school; 8-12 years, high school; and >13 years, college/university degree), and affinity for music (a 5-point scale: 1, 2, 3, 4, and 5 hours, measuring the length of time spent a day listening to music).

Data will be recorded by a single physician who will remain at the bedside throughout each session. Data will be analyzed in a blinded fashion another researcher who will be unaware of treatment allocations.

Power Analysis:

To achieve a power of 0.8 at α = 0.05 and one-tailed with a medium effect size of 0.610 and a medium correlation (r = 0.50) among two repeated measures using the F-test, a sample size of 30 mother-infant dyads will be needed.

ELIGIBILITY:
Inclusion criteria clinically stable infants

* postmenstrual age <37 weeks
* normal hearing confirmed by measurement of distortion product otoacoustic emission (DPOAE).

Exclusion criteria

* observed hyperresponsiveness to live music
* congenital anomaly that mainly affects hearing
* medication intake (phenobarbital, furosemide, gentamycin) that might interfere with the reaction to musical stimuli
* brain anomalies associated with neurological disorders (grade 3-4 intraventricular hemorrhage, periventricular leukomalacia).

Maternal inclusion criteria

* ability to hear
* literary ability to read and answer an anxiety questionnaire

Maternal exclusion criteria

* signs or medical history of postpartum depression

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduced Heart Rate | 30 minutes
Reduced respiratory rate | 30 minutes

SECONDARY OUTCOMES:
Als' Behavioral Score | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- NICU, Kfar Saba, Israel

REFERENCES:
- [Background] Hodges AL, Wilson LL. Effects of music therapy on preterm infants in the neonatal intensive care unit. Altern Ther Health Med. 2010 Sep-Oct;16(5):72-3. No abstract available. PMID 20882735
- [Result] Schlez A, Litmanovitz I, Bauer S, Dolfin T, Regev R, Arnon S. Combining kangaroo care and live harp music therapy in the neonatal intensive care unit setting. Isr Med Assoc J. 2011 Jun;13(6):354-8. PMID 21809733
- [Result] Olischar M, Shoemark H, Holton T, Weninger M, Hunt RW. The influence of music on aEEG activity in neurologically healthy newborns >/=32 weeks' gestational age. Acta Paediatr. 2011 May;100(5):670-5. doi: 10.1111/j.1651-2227.2011.02171.x. Epub 2011 Mar 1. PMID 21261705